CLINICAL TRIAL: NCT04836559
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-40411813 as Adjunctive Therapy in Subjects With Focal Onset Seizures With Suboptimal Response to Levetiracetam or Brivaracetam
Brief Title: A Study to Investigate JNJ-40411813 in Combination With Levetiracetam or Brivaracetam in Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108943; 40411813EPY2001 (Other: Janssen Research & Development, LLC); 2020-003698-24 (EudraCT Number)
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Focal Onset Seizures
MeSH Terms: conditions — Seizures | interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-40411813 (Experimental): Participants will receive JNJ-40411813 twice a day (bid) up to 12 weeks in double blind period. Up to 3 different doses (low, medium, high) of JNJ-40411813 will be administered in this study. Participants will also receive concomitant anti-epileptic drugs (AEDs) one of which must include levetiracetam or brivaracetam. Immediately after the last study drug intake by the participants in the double-blind period, participants will enter into a 2-year open label extension (OLE) period and continue receiving JNJ-40411813 as well as the AEDs during OLE period.
  Interventions: Drug: JNJ-40411813
- Placebo (Placebo Comparator): Participants will receive JNJ-40411813 matching placebo (bid) up to 12 weeks. Participants will also receive concomitant AEDs one of which must include levetiracetam or brivaracetam during double blind period. Participants who had been receiving placebo in double blind period will start with the JNJ-40411813 dose in the OLE period.
  Interventions: Drug: JNJ-40411813; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-40411813 — JNJ-40411813 will be administered orally.
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of up to 3 dose levels of adjunctive JNJ-40411813 compared to placebo based on the time to baseline monthly seizure count in participants with focal onset seizures who are receiving levetiracetam or brivaracetam and up to 3 other anti-epileptic drugs (AEDs) (double-blind treatment period) and to evaluate the long-term efficacy and safety of adjunctive therapy with JNJ-40411813 in participants with epilepsy (open-label extension [OLE] period).

DETAILED DESCRIPTION:
JNJ-40411813 is a positive allosteric modulator (PAM) of the metabotropic glutamate receptor-2 (mGlu2), which is abundantly expressed in the forebrain and cerebellum. The mGlu2 receptor functions as a presynaptic auto-receptor that, upon activation, decreases the release of the excitatory neurotransmitter glutamate. Positive allosteric modulation of a receptor will result in the direct enhancement of the agonist-induced signal while PAMs themselves have generally no or low intrinsic activity at the receptor. The net effect of JNJ-40411813 is hypothesized to be a normalization of hyper-glutamatergic transmission. JNJ-40411813 is being evaluated for the treatment of disorders of the central nervous systems (CNS), such as epilepsy, and has been evaluated in schizophrenia and anxious depression. This study will consist of 1 to a maximum of 3 cohorts. In each cohort, for each participant the study consists of a screening period (up to minus [-] 8 weeks), an 8-week prospective pretreatment baseline period, an up to 12-week double-blind treatment period and a 2-year OLE period or a follow-up telephone visit 2 weeks after the last dose of study intervention. Safety assessments including physical and neurological examination, vital signs, 12 lead electrocardiogram (ECG), clinical chemistry, hematology, and urinalysis will be performed. The total maximal duration of the study is up to 2 years and 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 35 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2). Minimum body weight should be 40-kilogram (kg)
* Established diagnosis of focal epilepsy, for at least 1 year using the International League Against Epilepsy (ILAE) criteria. Participants should not be enrolled if they are known to have had fewer than 3 or more than 100 seizures in any monthly period in the past 6 months. It is preferred that participants have experience in maintaining a seizure e-diary
* Must have had a neuroimaging procedure within 10 years, including a computed tomography (CT) scan or magnetic resonance imaging (MRI), that excluded a progressive neurologic disorder; these procedures may be performed within the 8-week baseline period
* Cohort 1: Current treatment with at least 1 and up to 4 anti-epileptic drugs (AEDs) (including levetiracetam), administered at stable dosage(s) for at least 1 month before screening, and no new AEDs added for the previous 2 months; these AEDs must remain unchanged throughout the pretreatment and double-blind treatment periods (with the exception of dosage reductions of concomitant AEDs because of suspected elevated AED levels or side effects) Cohort 2 and beyond: Current treatment with at least 1 and up to 4 AEDs (including levetiracetam or brivaracetam), administered at the appropriate dosage(s) and for a sufficient treatment period before screening. These AEDs must remain unchanged throughout the pretreatment and double-blind treatment periods (with the exception of dosage reductions of concomitant AEDs because of suspected elevated AED levels or side effects). Important note: screening of participants receiving brivaracetam will start when enrolling for Cohort 2
* Currently showing inadequate response to levetiracetam, administered at the appropriate dosage(s) and for a sufficient treatment period, based on the judgment of the investigator
* Healthy based on clinical laboratory tests, physical examination, medical history, vital signs, and 12-lead ECG
* Men or women between 18 and 69 years old

Exclusion Criteria:

* Have a generalized epileptic syndrome
* Diagnosis of Lennox-Gastaut Syndrome
* Currently experiencing seizures that cannot be counted accurately
* History of any current or past nonepileptic seizures, including psychogenic seizures
* Known allergies, hypersensitivity, or intolerance to placebo, JNJ-40411813 or its excipients
* Current treatment with vagus nerve stimulation, deep brain and cortical stimulation for 1 year or less
* Planned epilepsy surgery within the next 6 months or completed epilepsy surgery less than (<) 6 months ago
* Current treatment with vigabatrin
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Current or past (within the past year) major psychotic disorder, such as schizophrenia, bipolar disorder, or other psychotic conditions, recent (within the past 6 months) interictal psychosis, and major depressive disorder (MDD) with psychotic features
* Exacerbation of MDD within the past 6 months; antidepressant use is allowed
* Has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 4 (active suicidal ideation with some intent to act, without specific plan) or 5 (active suicidal ideation with specific plan and intent) for ideation on the Columbia Suicide Severity Rating Scale (C-SSRS), or a history of suicidal behavior within the past 1 year, as validated by the CSSRS at screening
* Has a history of at least mild drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria within 1 year before Screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (69):
- United States (7):
  - Tucson Neuroscience Research, Tucson, Arizona
  - Research Institution of Orlando, LLC, Orlando, Florida
  - Accel Research Sites, Port Orange, Florida
  - Maine Medical Center, Scarborough, Maine
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Belgium (6):
  - AZ Sint-Jan, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Antwerpen, Edegem
  - Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU UCL Namur - Site Godinne, Yvoir
- Germany (7):
  - Vivantes Humboldt Klinikum, Berlin
  - Krankenhaus Mara - Bethel, Bielefeld
  - Universitatsklinikum Bonn, Bonn
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Diakonie Kork - Epilepsiezentrum, Kehl-Kork
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
- Poland (17):
  - Centrum Medyczne Neuromed Sp z o. o., Bydgoszcz
  - Copernicus Podmiot Leczniczy Sp. z o.o, Gdansk
  - MA LEK AM Maciejowscy Spolka Cywilna Centrum Terapii SM, Katowice
  - NEURO MEDIC Janusz Zbrojkiewicz Poradnia Wielospecjalistyczna, Katowice
  - NZOZ Wielospecjalistyczna Poradnia Lekarska 'Synapsis', Katowice
  - Specjalistyczne Gabinety Lekarskie, Krakow
  - Centrum Leczenia Padaczki i Migreny NZOZ, Krakow
  - Centrum Opieki Zdrowotnej Orkan Med Stec Michalska sj, Ksawerów
  - Clinical Best Solutions Sp. z o.o., Sp. K., Lublin
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - NZOZ NEURO KARD Ilkowski i Partnerzy Sp Partnerska Lekarzy, Poznan
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Neurosphera, Warsaw
  - Institute of Psychiatry and Neurology, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - ProNeuro Centrum Medyczne, Żory
- Russia (10):
  - Republic Clinical Hospital, Kazan'
  - Research Medical Center Your Health, Kazan'
  - Specialized clinical psychiatric hospital #1, Krasnodar
  - Clinical City Hospital #1, Moscow
  - Nizny Novgorod clinical psychiatric hospital 1, Nizny Novgorod
  - Psychoneurological Dispensary of Frunzensky District, Saint Petersburg
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Yaroslavl State Medical University, Yaroslavl
- South Korea (6):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hosp. Del Mar, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Centro Neurologia Avanzada Sevilla, Seville
  - Hosp. Mutua Terrassa, Terrassa
  - Centro de Inv. Avanzada Neurociencias, Zaragoza
- Ukraine (7):
  - Ce 'Dnipropetrovsk Regional Clinical Hospital N.A. Mechnikov' of Dnipropetrovsk Rc, Dnipro
  - Medical Center of Private Enterprise Neuron, Kharkiv
  - Cnce of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Mnpe 'Regional Clinical Psychiatric Hospital of Kirovohrad Regional Council', Nove Settlement
  - Mnce 'Ternopil Regional Clinical Psychoneurology Hospital' of Trb, Ternopil
  - Llc Diamed Medical Center, Uzhhorod
  - Cnpe 'Vinnytsia Regional Clinical Psycho-Neurological Hospital N.A. Ac. O.I. Yushchenko' of Vrc, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diagnosis of focal onset seizures and receiving levetiracetam or brivaracetam and up to 3 other anti-epileptic drugs (AEDs) were enrolled in study. Study consisted of cohort 1 and 2. In each cohort, participants were stratified into two groups: participants treated with a CYP3A4 enzyme inducing anti-epileptic drugs (EIAED [induced participants]) and those not treated with a CYP3A4 EIAED (non-induced participants).
Pre-assignment Details: PK sets: randomized participants who received at least (>=)1 dose of JNJ-40411813 and had >=1 valid blood sample drawn for PK analysis and excluded samples with below lower limit of quantification or with inconsistent date/time or with previous dose date/time incomplete or samples with concentration <10 nanograms per milliliter. Safety set: randomized participants who received >=1 dose of JNJ-40411813/placebo. Due to inclusion/exclusion criteria difference, PK set count differed from safety set.
Groups:
- DB: Cohort 1: Placebo: During double-blind (DB) period, participants were randomized to receive placebo matching to JNJ-40411813 tablet orally twice a day (BID) from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the open-label extension (OLE) period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 1: JNJ-40411813: During DB period, participants were randomized to receive JNJ-40411813 100 milligrams (mg) or 50 mg tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants treated with EIAEDs (induced) received 100 mg of JNJ-40411813 and participants not treated with EIAEDs (non-induced) received 50 mg of JNJ-40411813. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continued DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: Placebo: During DB period, participants were randomized to receive placebo matching to JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: JNJ-40411813: During DB period, participants were randomized to receive JNJ-40411813 200 mg or 100 mg tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants treated with EIAEDs (induced) received 200 mg of JNJ-40411813 and participants not treated with EIAEDs (non-induced) received 100 mg of JNJ-40411813. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study drug due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- OLE: Cohort 1: Placebo Followed by JNJ-40411813: During OLE period, cohort 1 participants who had received placebo during the DB period received JNJ-40411813 100 mg or 50 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) received JNJ-40411813 100 mg, and non-induced participants (without EIAEDs) received JNJ-40411813 50 mg. The dose could be increased at the second visit (Month 1) to 200 mg of JNJ-40411813 BID for induced participants (with EIAEDs) and 100 mg of JNJ-40411813 BID for non-induced participants (without EIAEDs).
- OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813: During OLE period, cohort 1 participants who had received JNJ-40411813 during the DB period continued to receive JNJ-40411813 100 mg or 50 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) received JNJ-40411813 100 mg, and non-induced participants (without EIAEDs) received JNJ-40411813 50 mg. The dose could be increased at the second visit (Month 1) to 200 mg of JNJ-40411813 BID for induced participants (with EIAEDs) and 100 mg of JNJ-40411813 BID for non-induced participants (without EIAEDs).
- OLE: Cohort 2: Placebo Followed by JNJ-40411813: During the OLE period, cohort 2 participants who had received placebo during the DB period received JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Participants started with JNJ-40411813 100 mg BID. Induced participants (with EIAEDs) had their dose increased to JNJ-40411813 200 mg BID on Day 8 of the OLE. Non-induced participants (without EIAEDs) continued with JNJ-40411813 100 mg BID.
- OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813: During OLE period, cohort 2 participants who had received JNJ-40411813 during the DB period continued to receive JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Participants started with JNJ-40411813 100 mg BID. Induced participants (with EIAEDs) had their dose increased to JNJ-40411813 200 mg BID on Day 8 of the OLE. Non-induced participants (without EIAEDs) continued with JNJ-40411813 100 mg BID.
Period: Double Blind Period (Day 1 to Day 85)
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813 | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Started | 20 | 40 | 9 | 41 | 0 | 0 | 0 | 0
Full Analysis Set (All randomized participants assigned to receive study intervention and had both baseline and postbaseline seizure data.) | 20 | 40 | 9 | 40 | 0 | 0 | 0 | 0
Subjects Treated With EIAED | 11 | 22 | 6 | 24 | 0 | 0 | 0 | 0
Subjects Not Treated With EIAED | 9 | 18 | 3 | 17 | 0 | 0 | 0 | 0
Completed | 18 | 35 | 7 | 36 | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized by Mistake With Study Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: OLE Period (Day 1 of OLE up to 2 Years)
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813 | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Started | 0 | 0 | 0 | 0 | 12 | 23 | 7 | 31
Participants Treated With EIAED | 0 | 0 | 0 | 0 | 6 | 15 | 4 | 19
Participants Not Treated With EIAED | 0 | 0 | 0 | 0 | 6 | 8 | 3 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 23 | 7 | 31
Not completed — Sponsor's Decision | 0 | 0 | 0 | 0 | 7 | 14 | 4 | 24
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2
Not completed — No Longer Clinically Benefitting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813 | Total
Number analyzed (Participants) | 20 | 40 | 9 | 41 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (12.55) | 37.5 (12.40) | 39.7 (10.84) | 41.3 (11.47) | 39.8 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 17 | 5 | 23 | 50
  Male | 15 | 23 | 4 | 18 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 5 | 12
  Not Hispanic or Latino | 19 | 37 | 5 | 36 | 97
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 5 | 11 | 0 | 10 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 29 | 8 | 30 | 82
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 2 | 2
  Germany | 1 | 2 | 1 | 3 | 7
  Poland | 7 | 9 | 3 | 18 | 37
  Russian Federation | 2 | 7 | 0 | 0 | 9
  Korea, South | 5 | 11 | 0 | 9 | 25
  Spain | 0 | 3 | 4 | 7 | 14
  Ukraine | 2 | 5 | 0 | 0 | 7
  United States | 3 | 3 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 and 2: Time to Baseline Monthly Seizure Count up to the End of the 12-week Double-blind (DB) Treatment Period
Description: Time (in days) to baseline monthly seizure count was defined as the number of days until the participants cumulative seizure count during the DB period was equal to their baseline monthly seizure count. The baseline monthly seizure count was defined as the number of observable focal onset seizures occurred during the 8-week baseline period (Day -56 to -1), multiplied by 28/XBL, where XBL was the number of days comprising the participants baseline period. Observable focal onset seizures included focal aware seizures with motor signs, focal impaired awareness seizures and focal to bilateral tonic-clonic seizures. Focal aware seizures without motor signs, myoclonic, or other generalized seizures was not counted towards baseline monthly seizure count. Cluster seizures were counted as a single seizure. Kaplan-Meier method was used for the analysis.
Time Frame: From DB period Day 1 up to Day 85
Population: Full analysis set (FAS) included all randomized participants assigned to receive study intervention and had both baseline and postbaseline seizure data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 40
Days | 32 [28 to 37] | 34 [27 to 48] | 29 [22 to 69] | 38 [28 to 48]
Statistical Analysis 1: Comparison: DB: Cohort 1: Placebo vs DB: Cohort 1: JNJ-40411813; Test type: Superiority; p = 0.3571, t-test, 1 sided; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.41 to 1.38]
Statistical Analysis 2: Comparison: DB: Cohort 2: Placebo vs DB: Cohort 2: JNJ-40411813; Test type: Superiority; p = 0.6306, t-test, 1 sided; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.40 to 1.75]

2. Secondary Outcome: Cohort 1 and 2: Percent Reduction in the Open Label Extension (OLE) Period Monthly Seizure Rate
Description: The percent reduction in the OLE monthly seizure rate was defined as 100*(baseline monthly seizure count minus OLE monthly seizure count) divided by (baseline monthly seizure count). The OLE monthly seizure count was defined as the total number of observable focal onset seizures occurred during the OLE period, multiplied by 28/XOLE, where XOLE was the number of days comprising the OLE. A positive percentage change in the OLE monthly seizure count indicated improvement. Observable seizures included focal aware seizures with motor signs, focal impaired awareness seizures and focal to bilateral tonic-clonic seizures. Focal aware seizures without motor signs, myoclonic, or other generalized seizures was not counted towards baseline monthly seizure count. Cluster seizures were counted as a single seizure.
Time Frame: From OLE baseline (Day 1 of OLE) up to 24 months after start of OLE (the actual OLE starting time varied for each participant)
Population: Full analysis set: open-label extension (FASOLE) analysis set included all FAS participants who received at least 1 dose of study intervention in the OLE period.
Measure: Median (Inter-Quartile Range); unit: Percent change (reduction)
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 12 | 23 | 7 | 31
Percent change (reduction) | 39.9 [14.3 to 64.1] | 49.1 [-1.5 to 77.1] | 29.1 [22.6 to 76.6] | 52.1 [-3.7 to 85.0]

3. Secondary Outcome: Cohort 1 and 2: Number of Participants With Seizure Freedom at the End of OLE Period
Description: Number of participants with seizure freedom at the end of OLE period was reported. Seizure freedom was defined as having no seizures over the complete OLE study period.
Time Frame: as for outcome 2
Population: FASOLE analysis set included all FAS participants who received at least 1 dose of study intervention in the OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 12 | 23 | 7 | 31
Participants | 1 [14.3 to 64.1] | 0 [-1.5 to 77.1] | 0 [22.6 to 76.6] | 3 [-3.7 to 85.0]

4. Secondary Outcome: Cohort 1 and 2: Number of Participants With at Least 50 Percent (%) Reduction (Response) in the OLE Monthly Seizure Count
Description: Number of participants having at least a 50% reduction in the monthly seizure rate (response) during the OLE study period was reported.
Time Frame: as for outcome 2
Population: FASOLE analysis set included all FAS participants who received at least 1 dose of study intervention in the OLE period.
Measure: Count of Participants; unit: Participants
Groups:
- OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813: During OLE period, cohort 1 participants who had received JNJ-40411813 during the DB period continued to receive JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) received JNJ-40411813 100 mg BID, and non-induced participants (without EIAEDs) received JNJ-40411813 50 mg BID. The dose could be increased at the second visit (Month 1) to 200 mg of JNJ-40411813 BID for induced participants (with EIAEDs) and 100 mg of JNJ-40411813 BID for non-induced participants (without EIAEDs).
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 12 | 23 | 7 | 31
Participants | 5 | 11 | 3 | 16

5. Secondary Outcome: OLE Period: Cohort 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TEAEs and TESAEs were reported. An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A serious AE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product, or was medically important. TEAE/TESAE was defined as any AE/SAE occurred at or after the initial administration of study intervention through the day of last dose plus 5 days. TEAEs included serious and non-serious events.
Time Frame: From OLE baseline (Day 1 of OLE) up to 5 days after last dose of OLE period (5 days + 24 months after start of OLE) (the actual OLE starting time varied for each participant)
Population: Safety open label extension (SAFOLE) analysis set included all randomized participants who received at least 1 dose of study intervention in the OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 12 | 23 | 7 | 31
Participants
  TEAEs | 6 | 16 | 6 | 17
  TESAEs | 0 | 5 | 0 | 1

6. Secondary Outcome: OLE Period: Cohort 1 and 2: Number of Participants With Treatment-emergent (TE) Clinically Important Changes in Vital Signs
Description: TE clinically important changes in vital signs (VS) were pulse rate (PR) greater than (>)100 beats per min [bpm] and with >30bpm increase from baseline (BL), PR less than (<)50 bpm and with >20bpm decrease from BL, systolic blood pressure (SBP) >140 millimeters of mercury (mmHg) and with >40mm Hg increase from BL, SBP <90mmHg and with >30mmHg decrease from BL), diastolic blood pressure (DBP) >90mmHg and with >30mmHg increase from BL, DBP <50mmHg and with >20 mmHg decrease from BL, and temperature >38 degree Celsius(C) and with greater than or equal to (>=)1degree C increase from BL. TE: post BL value was above upper limit and BL value was below upper limit (example: Normal or Low). Same applied to post BL value being below lower limit with BL value being above lower limit (example: Normal or High). TEVS: VS which occurred as at or after initial administration of study intervention through last dose plus 5 days. Only categories in which at least 1 participant had data were reported.
Time Frame: From OLE baseline (Day 1 of OLE) up to 24 months + 5 days after start of OLE (the actual OLE starting time varied for each participant)
Population: SAFOLE analysis set included all randomized participants who received at least 1 dose of study intervention in the OLE period. Here 'N' (overall number of participants analyzed) refers to the number of participants with at least 1 postbaseline value for the specified vital sign parameter and 'n' (number analyzed) refers to number of participants evaluable at specified parameter. n=0 indicates that there was no evaluable participant for specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 0 | 1 | 0 | 1
Participants
  PR>100bpm with >30bpm increase from BL |  | 1 |  | 1
  SBP >140 mm Hg and with >40 mm Hg increase from BL: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP >140 mm Hg and with >40 mm Hg increase from BL |  | 1 |  |
  DBP >90 mm Hg, with >30 mm Hg increase from BL: number analyzed (Participants) | 0 | 1 | 0 | 0
  DBP >90 mm Hg, with >30 mm Hg increase from BL |  | 1 |  |

7. Secondary Outcome: OLE Period: Cohort 1 and 2: Number of Participants With Changes in Laboratory Assessments Recorded as TEAE
Description: Number of participants with changes in laboratory assessments recorded as TEAE were reported. Laboratory assessments included clinical chemistry, hematology and urinalysis. Postbaseline abnormalities were compared with baseline values: if postbaseline value exceeding the upper limit (with baseline below upper limit) or falling below the lower limit (with baseline above lower limit) was considered treatment-emergent (TE); if baseline values were missing then any postbaseline abnormality was considered TE. TEAE was defined as any AE occurring at or after the initial administration of study intervention through the day of last dose plus 5 days.
Time Frame: From OLE baseline (Day 1 of OLE) up to 24 months + 5 days after start of OLE (the actual OLE starting time varied for each subject)
Population: SAFOLE analysis set included all randomized participants who received at least 1 dose of study intervention in the OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
Number analyzed (Participants) | 12 | 23 | 7 | 31
Participants
  Chemistry | 2 | 4 | 0 | 2
  Hematology | 0 | 1 | 0 | 1
  Urinalysis | 0 | 2 | 0 | 0

8. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TEAEs and TESAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A serious AE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product, or was medically important. TEAE/TESAE was defined as any AE/SAE occurred at or after the initial administration of study intervention through the day of last dose plus 5 days. TEAEs included serious and non-serious events.
Time Frame: From DB period start (Day 1) up to 5 days after last dose of DB period (up to Day 90)
Population: Safety analysis set (SAF) included all randomized participants who received at least 1 dose of JNJ-40411813 or placebo in the double-blind period.
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 41
Participants
  TEAEs | 7 | 22 | 8 | 24
  TESAEs | 0 | 1 | 1 | 2

9. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Number of Participants With Treatment-emergent Clinically Important Changes in Vital Signs
Description: Treatment-emergent clinically important changes in vital signs defined as PR >100 bpm and with >30 bpm increase from baseline, PR <50 bpm and with >20 bpm decrease from baseline, SBP >140 mm Hg and with >40 mm Hg increase from baseline, SBP <90 mm Hg and with >30 mm Hg decrease from baseline, DBP >90 mm Hg and with >30 mm Hg increase from baseline, DBP <50 mm Hg and with >20 mm Hg decrease from baseline, temperature >38 degree C and with >=1 degree C increase from baseline. TE clinically important changes: if postbaseline value was above upper limit and baseline value was below upper limit (example: Normal or Low). Same applied to postbaseline value being below lower limit with baseline value being above lower limit (example: Normal or High). Only those categories in which at least 1 participant had data were reported in this outcome measure. TE vital signs included vital signs which occurred as at or after initial administration of study intervention through last dose plus 5 days.
Time Frame: From DB period start (Day 1) up to 5 days after last dose of DB period (up to Day 90)
Population: Safety analysis set included all randomized participants who received at least 1 dose of JNJ-40411813 or placebo in the double-blind period. Here 'N' (overall number of participants analyzed) refers to the number of participants with at least 1 postbaseline value for the specified vital sign parameter and 'n' (number analyzed) refers to number of participants evaluable at specified parameter. n=0 indicates that there was no evaluable participant for specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 1 | 1 | 0 | 2
Participants
  PR >100 bpm, >30 bpm increase from BL: number analyzed (Participants) | 0 | 1 | 0 | 2
  PR >100 bpm, >30 bpm increase from BL |  | 1 |  | 2
  SBP >140 mm Hg; with >40 mm Hg increase from BL: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP >140 mm Hg; with >40 mm Hg increase from BL |  | 1 |  |
  DBP >90 mm Hg and with >30 mm Hg increase from BL: number analyzed (Participants) | 1 | 0 | 0 | 0
  DBP >90 mm Hg and with >30 mm Hg increase from BL | 1 |  |  |

10. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Number of Participants With Treatment-emergent Clinically Important Changes in Electrocardiogram (ECG)
Description: The ECG parameters analyzed: heart rate, PR interval, RR interval, QRS interval, QT interval, and corrected QT (QTc) interval using the correction methods: Bazett's formula (QTcB), Fridericia's formula (QTcF). TE clinically important changes ECG values (relative to baseline) were defined as heart rate (bpm): <45 and >100; PR interval (millisecond [msec]): <120 and >200; QRS interval (msec): >120; QTc (msec): >470 in women and >450 in men. TE was concluded if the postbaseline value was above the upper limit and the baseline value was below the upper limit (example: Normal or Low). The same applied to the postbaseline value being below the lower limit with the baseline value being above the lower limit (example: Normal or High). TE ECGs: clinically important ECGs which occurred as at or after initial administration of study intervention through last dose plus 5 days. Only categories in which at least 1 participant had data were reported in this outcome measure.
Time Frame: From DB period start (Day 1) up to 5 days after last dose of DB period (up to Day 90)
Population: Safety analysis set included all randomized participants who received at least 1 dose of JNJ-40411813 or placebo in the double-blind period. Here 'n' (number analyzed) refers to number of participants with at least 1 postbaseline value for the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 41
Participants
  PR Interval (<120 msec): number analyzed (Participants) | 19 | 40 | 9 | 40
  PR Interval (<120 msec) | 1 | 2 | 0 | 2
  PR Interval (>200 msec): number analyzed (Participants) | 19 | 40 | 9 | 40
  PR Interval (>200 msec) | 0 | 2 | 1 | 2
  QRS Duration (>120 msec): number analyzed (Participants) | 19 | 40 | 9 | 40
  QRS Duration (>120 msec) | 0 | 2 | 0 | 1
  QTcB Interval (Female) (>470 msec): number analyzed (Participants) | 5 | 17 | 5 | 23
  QTcB Interval (Female) (>470 msec) | 1 | 0 | 0 | 0
  QTcB Interval (male) (>450 msec): number analyzed (Participants) | 14 | 23 | 4 | 17
  QTcB Interval (male) (>450 msec) | 0 | 1 | 0 | 2
  QTcF Interval (male) (>450 msec): number analyzed (Participants) | 14 | 23 | 4 | 17
  QTcF Interval (male) (>450 msec) | 0 | 0 | 0 | 1
  Heart Rate >100 beats/min: number analyzed (Participants) | 19 | 40 | 9 | 40
  Heart Rate >100 beats/min | 0 | 0 | 0 | 1

11. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Number of Participants With Changes in Laboratory Assessments Recorded as TEAE
Description: as for outcome 7
Time Frame: From DB period start (Day 1) up to 5 days after last dose of DB period (up to Day 90)
Population: Safety analysis set included all randomized participants who received at least 1 dose of JNJ-40411813 or placebo in the double-blind period.
Measure: Count of Participants; unit: Participants
Groups:
- DB: Cohort 1: Placebo: During double-blind (DB) period, participants were randomized to receive placebo matching to JNJ-40411813 tablet orally twice a day (BID) from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the open-label extension (OLE) period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 1: JNJ-40411813: During DB period, participants were randomized to receive JNJ-40411813 100 milligrams (mg) or 50 mg tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants treated with EIAEDs (induced) received 100 mg JNJ-40411813 and participants not treated with EIAEDs (non-induced) received 50 mg JNJ-40411813. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continued DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: Placebo: During DB period, participants were randomized to receive placebo matching to JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study visit for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: JNJ-40411813: During DB period, participants were randomized to receive JNJ-40411813 200 mg or 100 mg tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants treated with EIAEDs (induced) received 200 mg JNJ-40411813 and participants not treated with EIAEDs (non-induced) received 100 mg JNJ-40411813. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study drug due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 41
Participants
  Chemistry | 0 | 1 | 0 | 1
  Hematology | 0 | 0 | 0 | 1
  Urinalysis | 0 | 0 | 1 | 0

12. Secondary Outcome: Cohort 1 and 2: Percent Reduction in the Double-blind Period Monthly Seizure Rate
Description: The percent reduction in the DB monthly seizure rate was defined as 100*(baseline monthly seizure count minus DB monthly seizure count) divided by (baseline monthly seizure count). The DB monthly seizure count was defined as the total number of observable focal onset seizures occurring during the 12-week DB period, multiplied by 28/XDB, where XDB was the number of days comprising the DB period. A positive percentage change in the double-blind monthly seizure count indicates improvement. Observable focal onset seizures included focal aware seizures with motor signs, focal impaired awareness seizures and focal to bilateral tonic-clonic seizures. Focal aware seizures without motor signs, myoclonic, or other generalized seizures was not counted towards baseline monthly seizure count.
Time Frame: From DB period Day 1 up to Day 85
Population: FAS included all randomized participants assigned to receive study intervention and had both baseline and postbaseline seizure data.
Measure: Median (Inter-Quartile Range); unit: Percent change (reduction)
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 40
Percent change (reduction) | 23.0 [7.7 to 37.7] | 16.2 [-4.9 to 62.3] | 10.1 [-1.3 to 28.2] | 30.1 [-21.9 to 56.4]

13. Secondary Outcome: Cohort 1 and 2: Percentage of Participants With Seizure Freedom During Double-blind Period
Description: Percentage of participants with seizure freedom during DB period was reported. Seizure freedom was defined as having no seizures over the complete DB period.
Time Frame: From DB period Day 1 up to Day 85
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 40
Percentage of participants | 5.0 | 2.5 | 0.0 | 7.5

14. Secondary Outcome: Cohort 1 and 2: Percentage of Participants Who Achieved a More Than (>) 50 Percent (%) Reduction (Response) in Double-blind Monthly Seizure Count Relative to Baseline Monthly Seizure Count
Description: Percentage of participants who achieved a >50% reduction (response) in the DB monthly seizure count relative to baseline monthly seizure count during the DB period was reported. The baseline monthly seizure count was defined as the number of observable focal onset seizures occurred during the 8-week baseline period (Day -56 to -1), multiplied by 28/XBL, where XBL was the number of days comprising the participants baseline period. Observable focal onset seizures included focal aware seizures with motor signs, focal impaired awareness seizures and focal to bilateral tonic-clonic seizures. Focal aware seizures without motor signs, myoclonic, or other generalized seizures was not counted towards baseline monthly seizure count.
Time Frame: From DB period Day 1 up to Day 85
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813
Number analyzed (Participants) | 20 | 40 | 9 | 40
Percentage of participants | 15.0 | 32.5 | 22.2 | 30.0

15. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Plasma Concentration of JNJ-40411813 and Its Metabolites: M30, M45 and M47
Description: DB treatment period: Cohort 1 and 2: plasma concentration of JNJ-40411813 and its metabolites (M30, M45 and M47) were reported. The concentrations of JNJ-40411813 and its metabolites (M30, M45 and M47) were measured using a validated, specific, and sensitive liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) method. Data for this outcome measure was not planned to be collected and analyzed for Cohort 1 and 2 placebo arms. Here, 'n' (number analyzed)=number of participants evaluable at each specified category.
Time Frame: Day 1: 2 hours post-dose, Days 29: pre-dose and 1 hour post-dose, Day 57: pre-dose and Day 85: post-dose/Early withdrawal (EW)
Population: Pharmacokinetic (PK) set: all randomized participants who received at least 1 dose of JNJ-40411813 and had at least 1 valid blood sample drawn for PK analysis and excluded samples with below lower limit of quantification or samples with inconsistent date/time or samples with previous dose date/time incomplete or samples with concentration less than (<) 10 nanograms per milliliter (ng/mL).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- DB: Cohort 1: JNJ-40411813 Non-induced: During DB period, participants not treated with EIAEDs (non-induced) received 50 mg JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continued DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 1: JNJ-40411813 Induced: During DB period, participants treated with EIAEDs (induced) received 100 mg JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continued DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were follow-up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: JNJ-40411813 Non-induced: During DB period, participants not treated with EIAEDs (non-induced) received 100 mg JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were follow-up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: JNJ-40411813 Induced: During DB period, participants treated with EIAEDs (induced) received 200 mg JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform the end-of-study for DB period visit (last visit for last participant; Day 85) or enter the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were follow-up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
Arm/Group | DB: Cohort 1: JNJ-40411813 Non-induced | DB: Cohort 1: JNJ-40411813 Induced | DB: Cohort 2: JNJ-40411813 Non-induced | DB: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 18 | 22 | 17 | 22
Nanograms per milliliter
  JNJ: Day 1: 2 hours post-dose: number analyzed (Participants) | 16 | 21 | 16 | 19
  JNJ: Day 1: 2 hours post-dose | 228 (116) | 268 (139) | 212 (113) | 379 (192)
  JNJ: Day 29: pre-dose: number analyzed (Participants) | 15 | 18 | 15 | 19
  JNJ: Day 29: pre-dose | 272 (178) | 356 (192) | 506 (283) | 797 (412)
  JNJ: Day 29: 1 hour post-dose: number analyzed (Participants) | 15 | 18 | 15 | 21
  JNJ: Day 29: 1 hour post-dose | 403 (285) | 560 (281) | 633 (289) | 958 (465)
  JNJ: Day 57: pre-dose: number analyzed (Participants) | 15 | 15 | 11 | 12
  JNJ: Day 57: pre-dose | 276 (205) | 360 (187) | 516 (216) | 687 (248)
  JNJ: Day 85:post-dose/EW: number analyzed (Participants) | 14 | 19 | 13 | 15
  JNJ: Day 85:post-dose/EW | 354 (385) | 440 (343) | 515 (267) | 785 (394)
  M30: Day 1: 2 hours post-dose: number analyzed (Participants) | 14 | 20 | 14 | 16
  M30: Day 1: 2 hours post-dose | 20.8 (11.7) | 21.5 (15.5) | 12.6 (8.85) | 24.8 (20.4)
  M30: Day 29: pre-dose: number analyzed (Participants) | 13 | 16 | 14 | 16
  M30: Day 29: pre-dose | 326 (116) | 232 (109) | 294 (119) | 239 (100)
  M30: Day 29: 1 hour post-dose: number analyzed (Participants) | 13 | 18 | 14 | 18
  M30: Day 29: 1 hour post-dose | 295 (108) | 211 (105) | 275 (119) | 220 (116)
  M30: Day 57: pre-dose: number analyzed (Participants) | 16 | 15 | 13 | 12
  M30: Day 57: pre-dose | 291 (150) | 219 (108) | 289 (135) | 277 (111)
  M30: Day 85:post-dose/EW: number analyzed (Participants) | 15 | 19 | 12 | 14
  M30: Day 85:post-dose/EW | 299 (123) | 191 (122) | 248 (121) | 274 (93.7)
  M45: Day 1: 2 hours post-dose: number analyzed (Participants) | 15 | 20 | 14 | 16
  M45: Day 1: 2 hours post-dose | 58.9 (24.2) | 49.8 (31.0) | 45.1 (21.6) | 52.5 (22.5)
  M45: Day 29: pre-dose: number analyzed (Participants) | 13 | 16 | 14 | 16
  M45: Day 29: pre-dose | 107 (60.1) | 65.4 (45.7) | 122 (64.9) | 76.3 (35.2)
  M45: Day 29: 1 hour post-dose: number analyzed (Participants) | 13 | 18 | 14 | 18
  M45: Day 29: 1 hour post-dose | 106 (54.8) | 68.9 (36.3) | 115 (56.0) | 74.5 (28.4)
  M45: Day 57: pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 12
  M45: Day 57: pre-dose | 103 (55.7) | 63.6 (42.9) | 113 (56.8) | 76.0 (32.1)
  M45: Day 85: post-dose/EW: number analyzed (Participants) | 15 | 18 | 12 | 15
  M45: Day 85: post-dose/EW | 101 (57.9) | 62.3 (41.6) | 113 (64.2) | 73.5 (40.1)
  M47: Day 1: 2 hours post-dose: number analyzed (Participants) | 15 | 20 | 14 | 16
  M47: Day 1: 2 hours post-dose | 25.8 (14.0) | 34.7 (19.7) | 19.4 (10.5) | 36.8 (20.3)
  M47: Day 29: pre-dose: number analyzed (Participants) | 13 | 16 | 14 | 16
  M47: Day 29: pre-dose | 51.9 (36.1) | 63.7 (31.7) | 81.6 (41.5) | 93.8 (42.9)
  M47: Day 29: 1 hour post-dose: number analyzed (Participants) | 13 | 18 | 14 | 18
  M47: Day 29: 1 hour post-dose | 53.5 (30.5) | 69.7 (29.2) | 77.3 (36.4) | 90.1 (45.3)
  M47: Day 57: pre-dose: number analyzed (Participants) | 15 | 15 | 13 | 12
  M47: Day 57: pre-dose | 53.3 (47.5) | 61.7 (26.2) | 84.0 (41.7) | 94.3 (30.1)
  M47: Day 85: post-dose/EW: number analyzed (Participants) | 15 | 19 | 11 | 14
  M47: Day 85: post-dose/EW | 52.9 (58.8) | 60.2 (37.8) | 97.4 (27.8) | 100 (39.9)

16. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Plasma Concentration of AED: Levetiracetam
Description: DB treatment period: Cohort 1 and 2: plasma concentration of AED: levetiracetam were reported. The concentrations of levetiracetam were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Day 1: pre-dose and 2 hours post-dose, Day 29: pre-dose and 1 hour post-dose, Day 57: pre-dose and Day 85: post-dose/Early withdrawal
Population: PK set was used. Here, 'N' (overall number of participants analyzed)=number of participants evaluable for this OM; 'n' (number analyzed) = number of participants evaluable at each specified category.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- DB: Cohort 1: Placebo Non-induced: During DB period, participants not treated with EIAEDs (non-induced) received placebo matching to JNJ-40411813 tablet orally twice a day (BID) from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the open-label extension (OLE) period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 1: Placebo Induced: During DB period, participants treated with EIAEDs (induced) received placebo matching to JNJ-40411813 tablet orally twice a day (BID) from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the open-label extension (OLE) period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: Placebo Non-induced: During DB period, participants not treated with EIAEDs (non-induced) received placebo matching to JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- DB: Cohort 2: Placebo Induced: During DB period, participants treated with EIAEDs (induced) received placebo matching to JNJ-40411813 tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
Arm/Group | DB: Cohort 1: Placebo Non-induced | DB: Cohort 1: Placebo Induced | DB: Cohort 1: JNJ-40411813 Non-induced | DB: Cohort 1: JNJ-40411813 Induced | DB: Cohort 2: Placebo Non-induced | DB: Cohort 2: Placebo Induced | DB: Cohort 2: JNJ-40411813 Non-induced | DB: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 9 | 11 | 18 | 22 | 2 | 5 | 15 | 13
Nanograms per milliliter
  Day 1: pre-dose: number analyzed (Participants) | 6 | 9 | 13 | 17 | 2 | 5 | 14 | 11
  Day 1: pre-dose | 9443 (7244) | 9664 (4210) | 12719 (8734) | 10836 (7328) | 28950 (17748) | 23190 (26095) | 18844 (16282) | 11648 (11371)
  Day 1: 2 hours post-dose: number analyzed (Participants) | 9 | 10 | 17 | 19 | 2 | 5 | 15 | 11
  Day 1: 2 hours post-dose | 28926 (16762) | 28859 (15629) | 29782 (19304) | 21593 (13973) | 35450 (2475) | 27300 (11876) | 24638 (13687) | 22894 (13656)
  Day 29: pre-dose: number analyzed (Participants) | 8 | 9 | 13 | 16 | 1 | 3 | 15 | 9
  Day 29: pre-dose | 12420 (9133) | 16546 (13963) | 17583 (11268) | 8926 (6665) | 14400 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 7137 (247) | 17369 (11404) | 7651 (5505)
  Day 29: 1 hour post-dose: number analyzed (Participants) | 9 | 9 | 14 | 17 | 2 | 2 | 15 | 7
  Day 29: 1 hour post-dose | 27510 (24608) | 30999 (15392) | 28709 (14885) | 24383 (23858) | 28050 (18031) | 27950 (3041) | 22102 (14695) | 30887 (16987)
  Day 57: pre-dose: number analyzed (Participants) | 8 | 9 | 15 | 15 | 2 | 2 | 11 | 5
  Day 57: pre-dose | 14066 (11366) | 12992 (8088) | 12927 (6140) | 10403 (8785) | 9680 (10493) | 23900 (18950) | 18090 (11580) | 6786 (8500)
  Day 85: post-dose/EW: number analyzed (Participants) | 7 | 8 | 15 | 19 | 2 | 2 | 11 | 7
  Day 85: post-dose/EW | 19834 (19271) | 19671 (14617) | 23461 (20193) | 15451 (12004) | 40000 (2970) | 22950 (17466) | 20680 (15826) | 16053 (22950)

17. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Plasma Concentration of AED: Brivaracetam
Description: DB treatment period: Cohort 1 and 2: plasma concentration of AED: brivaracetam were reported. The concentrations of brivaracetam were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Day 1: pre-dose and 2 hours post-dose, Days 29: pre-dose and 1 hour post-dose, Day 57: pre-dose and Day 85: post-dose/Early withdrawal
Population: PK set was used for the analysis. Here, 'N' (overall number of participants analyzed)=number of participants evaluable for this OM; 'n' (number analyzed) = number of participants evaluable at each specified category. Here, N=0 signifies that no participant received brivaracetam; n=0 in arm 'DB: Cohort 2: Placebo Non-induced' at timepoint 'Day 57: pre-dose' signifies that no participant was available at specific visit and thus, no data was collected and analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | DB: Cohort 1: Placebo Non-induced | DB: Cohort 1: Placebo Induced | DB: Cohort 1: JNJ-40411813 Non-induced | DB: Cohort 1: JNJ-40411813 Induced | DB: Cohort 2: Placebo Non-induced | DB: Cohort 2: Placebo Induced | DB: Cohort 2: JNJ-40411813 Non-induced | DB: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 11
Nanograms per milliliter
  Day 1: pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 9
  Day 1: pre-dose |  |  |  |  | 556 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 1040 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 1604 (1394) | 838 (622)
  Day 1: 2 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 9
  Day 1: 2 hours post-dose |  |  |  |  | 2150 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2970 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2320 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2540 (1659)
  Day 29: pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 10
  Day 29: pre-dose |  |  |  |  | 750 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 991 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2495 (1619) | 734 (658)
  Day 29: 1 hour post-dose |  |  |  |  | 3230 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2950 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 3930 (85) | 2343 (1149)
  Day 57: pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 7
  Day 57: pre-dose |  |  |  |  |  | 1020 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 950 (284) | 709 (719)
  Day 85: post-dose/EW: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 8
  Day 85: post-dose/EW |  |  |  |  | 743 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 3330 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 2499 (2547) | 1258 (1444)

18. Secondary Outcome: DB Treatment Period: Cohort 1 and 2: Plasma Concentration of AED: Carbamazepine
Description: DB treatment period: Cohort 1 and 2: plasma concentration of AED: carbamazepine were reported. The concentrations of carbamazepine were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose: Day 1, Days 29, and Day 57
Population: PK set was used for the analysis. Here, 'N' (overall number of participants analyzed)=number of participants evaluable for this OM; 'n' (number analyzed) = number of participants evaluable at each specified category. Here, N=0 signifies that non-induced arms were not applicable to this outcome measure as carbamazepine itself is a CYP3A4-inducing AED.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | DB: Cohort 1: Placebo Non-induced | DB: Cohort 1: Placebo Induced | DB: Cohort 1: JNJ-40411813 Non-induced | DB: Cohort 1: JNJ-40411813 Induced | DB: Cohort 2: Placebo Non-induced | DB: Cohort 2: Placebo Induced | DB: Cohort 2: JNJ-40411813 Non-induced | DB: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 0 | 5 | 0 | 12 | 0 | 2 | 0 | 12
Nanograms per milliliter
  Day 1: pre-dose |  | 7618 (3305) |  | 5071 (3773) |  | 7450 (1966) |  | 7431 (1214)
  Day 29: pre-dose: number analyzed (Participants) | 0 | 4 | 0 | 9 | 0 | 2 | 0 | 10
  Day 29: pre-dose |  | 8270 (1481) |  | 4713 (4198) |  | 6990 (269) |  | 6476 (1895)
  Day 57: pre-dose: number analyzed (Participants) | 0 | 4 | 0 | 8 | 0 | 1 | 0 | 6
  Day 57: pre-dose |  | 7943 (1975) |  | 4526 (2765) |  | 6390 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. |  | 5573 (915)

19. Secondary Outcome: OLE Period: Cohort 1 and 2: Plasma Concentration of JNJ-40411813 and Its Metabolites: M30, M45 and M47
Description: OLE period: Cohort 1 and 2: plasma concentration of JNJ-40411813 and its metabolites (M30, M45 and M47) were reported. The concentrations of JNJ-40411813 and its metabolites (M30, M45 and M47) were measured using a validated, specific, and sensitive LC-MS/MS method. Data for this outcome measure was not planned to be collected and analyzed for Cohort 1 and 2 placebo arms. OLE baseline was Day 1 of OLE period.
Time Frame: Cohort 1:OLE visit 2 (1 month post OLE baseline[BL]), OLE visit 3 (2 months post OLE BL), OLE visit 4 to 7 (up to 1year post OLE BL);Cohort 2:OLE visit 2 (1 month post OLE BL), OLE visit 3 (2 months post OLE BL), OLE visit 4 to 5 (up to 1year post OLE BL)
Population: PK set was used for the analysis. Here, n=0 signifies that none of the participants were evaluable for assessment in the specified arm for specified time point. Here, 'n' (number analyzed)=number of participants evaluable at each specified category.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- OLE: Cohort 1: JNJ-40411813 Non-induced: During OLE period, cohort 1 non-induced participants (without EIAEDs) received JNJ-40411813 50 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. The dose could be increased at the second visit (Month 1) to 100 mg JNJ-40411813 BID.
- OLE: Cohort 1: JNJ-40411813 Induced: During OLE period, cohort 1 induced participants (with EIAEDs) received JNJ-40411813 100 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. The dose could be increased at the second visit (Month 1) to 200 mg JNJ-40411813 BID.
- OLE: Cohort 2: JNJ-40411813 Non-induced: During the OLE period, cohort 2 participants started with JNJ-40411813 100 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Non-induced participants (without EIAEDs) continued with JNJ-40411813 100 mg BID up to 2 years of OLE.
- OLE: Cohort 2: JNJ-40411813 Induced: During the OLE period, cohort 2 participants started with JNJ-40411813 100 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) had their dose increased to JNJ-40411813 200 mg BID on Day 8 up to 2 years of OLE.
Arm/Group | OLE: Cohort 1: JNJ-40411813 Non-induced | OLE: Cohort 1: JNJ-40411813 Induced | OLE: Cohort 2: JNJ-40411813 Non-induced | OLE: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 8 | 15 | 11 | 16
Nanograms per milliliter
  JNJ-40411813: OLE visit 2: number analyzed (Participants) | 8 | 14 | 11 | 16
  JNJ-40411813: OLE visit 2 | 272 (233) | 372 (241) | 524 (149) | 930 (370)
  JNJ-40411813: OLE visit 3: number analyzed (Participants) | 8 | 13 | 8 | 14
  JNJ-40411813: OLE visit 3 | 280 (217) | 333 (157) | 515 (172) | 993 (361)
  JNJ-40411813: OLE visit 4: number analyzed (Participants) | 6 | 12 | 4 | 11
  JNJ-40411813: OLE visit 4 | 311 (207) | 392 (288) | 539 (147) | 921 (464)
  JNJ-40411813: OLE visit 5: number analyzed (Participants) | 5 | 11 | 2 | 2
  JNJ-40411813: OLE visit 5 | 285 (241) | 315 (197) | 532 (105) | 1610 (255)
  JNJ-40411813: OLE visit 6: number analyzed (Participants) | 4 | 10 | 0 | 0
  JNJ-40411813: OLE visit 6 | 442 (493) | 349 (214) |  |
  JNJ-40411813: OLE visit 7: number analyzed (Participants) | 4 | 7 | 0 | 0
  JNJ-40411813: OLE visit 7 | 330 (252) | 385 (269) |  |
  M30: OLE visit 2: number analyzed (Participants) | 7 | 14 | 10 | 15
  M30: OLE visit 2 | 298 (91.3) | 225 (136) | 316 (129) | 249 (94.9)
  M30: OLE visit 3: number analyzed (Participants) | 8 | 14 | 8 | 14
  M30: OLE visit 3 | 293 (135) | 224 (172) | 356 (113) | 234 (73.7)
  M30: OLE visit 4: number analyzed (Participants) | 6 | 12 | 4 | 11
  M30: OLE visit 4 | 265 (120) | 263 (161) | 333 (125) | 251 (54.6)
  M30: OLE visit 5: number analyzed (Participants) | 5 | 11 | 2 | 2
  M30: OLE visit 5 | 301 (154) | 259 (169) | 349 (223) | 274 (65.1)
  M30: OLE visit 6: number analyzed (Participants) | 4 | 10 | 0 | 0
  M30: OLE visit 6 | 286 (91.8) | 236 (141) |  |
  M30: OLE visit 7: number analyzed (Participants) | 4 | 7 | 0 | 0
  M30: OLE visit 7 | 364 (64.7) | 265 (115) |  |
  M45: OLE visit 2: number analyzed (Participants) | 7 | 14 | 10 | 15
  M45: OLE visit 2 | 85.3 (37.8) | 57.7 (29.2) | 101 (34.9) | 87.4 (27.8)
  M45: OLE visit 3: number analyzed (Participants) | 8 | 13 | 8 | 14
  M45: OLE visit 3 | 93.8 (41.2) | 56.0 (28.0) | 101 (54.5) | 85.5 (29.0)
  M45: OLE visit 4: number analyzed (Participants) | 6 | 12 | 4 | 11
  M45: OLE visit 4 | 81.1 (40.9) | 64.0 (32.4) | 112 (77.0) | 84.0 (30.7)
  M45: OLE visit 5: number analyzed (Participants) | 5 | 11 | 2 | 2
  M45: OLE visit 5 | 75.7 (45.2) | 65.7 (38.0) | 89.2 (9.69) | 91.7 (6.22)
  M45: OLE visit 6: number analyzed (Participants) | 4 | 10 | 0 | 0
  M45: OLE visit 6 | 72.1 (49.8) | 61.6 (41.9) |  |
  M45: OLE visit 7: number analyzed (Participants) | 4 | 7 | 0 | 0
  M45: OLE visit 7 | 71.8 (51.9) | 59.3 (28.4) |  |
  M47: OLE visit 2: number analyzed (Participants) | 7 | 14 | 10 | 15
  M47: OLE visit 2 | 59.3 (71.0) | 58.0 (31.4) | 98.9 (34.6) | 107 (30.8)
  M47: OLE visit 3: number analyzed (Participants) | 8 | 13 | 8 | 14
  M47: OLE visit 3 | 52.8 (58.2) | 58.7 (24.5) | 81.7 (28.6) | 122 (45.4)
  M47: OLE visit 4: number analyzed (Participants) | 6 | 12 | 4 | 11
  M47: OLE visit 4 | 59.1 (66.0) | 65.6 (34.1) | 80.3 (12.4) | 118 (47.1)
  M47: OLE visit 5: number analyzed (Participants) | 5 | 11 | 2 | 2
  M47: OLE visit 5 | 62.8 (79.1) | 57.6 (25.1) | 78.0 (13.9) | 157 (58.0)
  M47: OLE visit 6: number analyzed (Participants) | 4 | 10 | 0 | 0
  M47: OLE visit 6 | 70.1 (90.8) | 66.9 (44.9) |  |
  M47: OLE visit 7: number analyzed (Participants) | 4 | 7 | 0 | 0
  M47: OLE visit 7 | 70.3 (80.7) | 69.8 (30.4) |  |

20. Secondary Outcome: OLE Period: Cohort 1 and 2: Plasma Concentration of AED: Levetiracetam
Description: OLE period: Cohort 1 and 2: plasma concentration of AED: levetiracetam were reported. The concentrations of levetiracetam were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: OLE visit 2: 1st month; OLE visit 3: 2nd month
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- OLE: Cohort 1: Placebo Followed by JNJ-40411813 Non-induced: During OLE period, cohort 1 non-induced participants (without EIAEDs) who had received placebo matched to JNJ-40411813 during the DB period received JNJ-40411813 50 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. The dose could be increased at the second visit (Month 1) to 100 mg of JNJ-40411813 BID for non-induced participants (without EIAEDs).
- OLE: Cohort 1: Placebo Followed by JNJ-40411813 Induced: During OLE period, cohort 1 induced participants (with EIAEDs) who had received placebo matched to JNJ-40411813 during the DB period received JNJ-40411813 100 mg BID along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. The dose could be increased at the second visit (Month 1) to 200 mg of JNJ-40411813 BID for induced participants (with EIAEDs).
- OLE: Cohort 2: Placebo Followed by JNJ-40411813 Non-induced: During the OLE period, cohort 2 non-induced participants (without EIAEDs) who had received placebo matched to JNJ-40411813 during the DB period received JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Participants started with JNJ-40411813 100 mg BID. Non-induced participants (without EIAEDs) continued with JNJ-40411813 100 mg BID.
- OLE: Cohort 2: Placebo Followed by JNJ-40411813 Induced: During the OLE period, cohort 2 induced participants (with EIAEDs) who had received placebo matched to JNJ-40411813 during the DB period received JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Participants started with JNJ-40411813 100 mg BID. Induced participants (with EIAEDs) had their dose increased to JNJ-40411813 200 mg BID on Day 8 of the OLE.
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 1: JNJ-40411813 Non-induced | OLE: Cohort 1: JNJ-40411813 Induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 2: JNJ-40411813 Non-induced | OLE: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 2 | 4 | 8 | 14 | 2 | 1 | 9 | 7
Nanograms per milliliter
  OLE visit 2: number analyzed (Participants) | 2 | 4 | 7 | 12 | 2 | 1 | 9 | 7
  OLE visit 2 | 12980 (6817) | 9752 (2937) | 15787 (6029) | 11719 (7661) | 15000 (849) | 7410 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 15406 (7870) | 11929 (13102)
  OLE visit 3: number analyzed (Participants) | 1 | 4 | 7 | 12 | 2 | 1 | 5 | 6
  OLE visit 3 | 10400 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 8310 (3019) | 15734 (7392) | 10643 (7986) | 12100 (1273) | 29100 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 13760 (4972) | 5068 (5040)

21. Secondary Outcome: OLE Period: Cohort 1 and 2: Plasma Concentration of AED: Brivaracetam
Description: OLE period: Cohort 1 and 2: plasma concentration of AED: brivaracetam were reported. The concentrations of brivaracetam were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: OLE visit 2: 1st month; OLE visit 3: 2nd month
Population: PK set was used. 'N' (overall number of participants analyzed)=number of participants evaluable for this OM; 'n' (number analyzed)=number of participants evaluable at each specified category. Cohort (C) 1: N=0=no participant received brivaracetam; C 2: N=0=no participant was available and thus, no data was collected and analyzed; n=0 in arm 'OLE: C 2: JNJ-40411813 Non-induced' timepoint 'OLE visit 3'= no participant was available at specific visit and thus, no data was collected and analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 1: JNJ-40411813 Non-induced | OLE: Cohort 1: JNJ-40411813 Induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 2: JNJ-40411813 Non-induced | OLE: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8
Nanograms per milliliter
  OLE visit 2 |  |  |  |  |  | 1030 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 611 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. | 834 (707)
  OLE visit 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
  OLE visit 3 |  |  |  |  |  | 1010 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. |  | 694 (746)

22. Secondary Outcome: OLE Period: Plasma Concentration of AED: Carbamazepine
Description: OLE period: Cohort 1 and 2: plasma concentration of AED: carbamazepine were reported. The concentrations of carbamazepine were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: OLE visit 2: 1st month; OLE visit 3: 2nd month
Population: PK set used. 'N' (overall number of participants analyzed)=number of participants evaluable for this OM; 'n' (number analyzed) = number of participants evaluable at each specified category. N=0 of all non-induced arms signifies that these arms were not applicable to this outcome measure as carbamazepine itself is a CYP3A4-inducing AED; For 'OLE: Cohort 2: Placebo Followed by JNJ-40411813 Induced' arm: N=0 signifies that no participant was available and thus, no data was collected and analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 1: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 1: JNJ-40411813 Non-induced | OLE: Cohort 1: JNJ-40411813 Induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Non-induced | OLE: Cohort 2: Placebo Followed by JNJ-40411813 Induced | OLE: Cohort 2: JNJ-40411813 Non-induced | OLE: Cohort 2: JNJ-40411813 Induced
Number analyzed (Participants) | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 5
Nanograms per milliliter
  OLE visit 2: number analyzed (Participants) | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 5
  OLE visit 2 |  | 5970 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. |  | 3780 (2604) |  |  |  | 6266 (1370)
  OLE visit 3: number analyzed (Participants) | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 4
  OLE visit 3 |  | 5780 (NA) — Here, 'NA' signifies that standard deviation could not be estimated as only 1 participant was analyzed. |  | 5814 (4617) |  |  |  | 6638 (1868)

ADVERSE EVENTS:
Time Frame: DB arms: From DB period start (Day 1) up to 5 days after last dose of DB period (up to Day 90); OLE arms: From OLE baseline (Day 1 of OLE) up to 24 months after start of OLE (the actual OLE starting time varied for each participant)
Description: DB period: SAF included all randomized participants who received at least 1 dose of JNJ-40411813 or placebo in the DB period. OLE period: SAFOLE analysis set included all randomized participants who received at least 1 dose of study intervention in the OLE period.
Groups:
- DB: Cohort 2: JNJ-40411813: During DB period, participants were randomized to receive JNJ-40411813 200 mg or 100 mg tablet orally BID from Day 1 up to Day 85 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) on Days 1, 29, and 57. Participants treated with EIAEDs (induced) received 200 mg of JNJ-40411813 and participants not treated with EIAEDs (non-induced) received 100 mg of JNJ-40411813. Participants were screened every 4 weeks for monthly seizure counts up to Week 12. Participants who had exceeded their pre-randomization monthly seizure count had the option to discontinue the study treatment due to lack of efficacy and perform the end-of-study/early withdrawal visit, continue DB treatment, or enter the OLE period. Participants who had not exceeded the pre-randomization seizure count continued the DB treatment period through Week 12 and had the option to perform DB period end-of-study visit (last visit for last participant; Day 85) or entered the OLE period. Participants who continued treatment to the end of the DB period (Week 12) and were not elected to participate in the OLE were followed up for safety up to 2 weeks after the last dose of study treatment (up to Week 14).
- OLE: Cohort 1: Placebo Followed by JNJ-40411813: During OLE period, cohort 1 participants who had received placebo during the DB period received JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) received JNJ-40411813 100 mg BID, and non-induced participants (without EIAEDs) received JNJ-40411813 50 mg BID. The dose could be increased at the second visit (Month 1) to 200 mg JNJ-40411813 BID for induced participants (with EIAEDs) and 100 mg JNJ-40411813 BID for non-induced participants (without EIAEDs).
- OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813: During OLE period, cohort 1 participants who had received JNJ-40411813 during the DB period continued to receive JNJ-40411813 along with previously prescribed AEDs (one of which must include levetiracetam or brivaracetam) from Day 1 of OLE up to 2 years. Induced participants (with EIAEDs) received JNJ-40411813 100 mg BID, and non-induced participants (without EIAEDs) received JNJ-40411813 50 mg BID. The dose could be increased at the second visit (Month1) to 200 mg JNJ-40411813 BID for induced participants (with EIAEDs) and 100 mg JNJ-40411813 BID for non-induced participants (without EIAEDs).
Arm/Group | DB: Cohort 1: Placebo | DB: Cohort 1: JNJ-40411813 | DB: Cohort 2: Placebo | DB: Cohort 2: JNJ-40411813 | OLE: Cohort 1: Placebo Followed by JNJ-40411813 | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 | OLE: Cohort 2: Placebo Followed by JNJ-40411813 | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/40 | 0/9 | 0/41 | 0/12 | 0/23 | 0/7 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/40 | 1/9 | 2/41 | 0/12 | 5/23 | 0/7 | 1/31
Other Adverse Events (participants affected / at risk) | 7/20 | 16/40 | 7/9 | 19/41 | 6/12 | 12/23 | 6/7 | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Cohort 1: Placebo (N=20) | DB: Cohort 1: JNJ-40411813 (N=40) | DB: Cohort 2: Placebo (N=9) | DB: Cohort 2: JNJ-40411813 (N=41) | OLE: Cohort 1: Placebo Followed by JNJ-40411813 (N=12) | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 (N=23) | OLE: Cohort 2: Placebo Followed by JNJ-40411813 (N=7) | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813 (N=31)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Change in Seizure Presentation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Status Epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Cohort 1: Placebo (N=20) | DB: Cohort 1: JNJ-40411813 (N=40) | DB: Cohort 2: Placebo (N=9) | DB: Cohort 2: JNJ-40411813 (N=41) | OLE: Cohort 1: Placebo Followed by JNJ-40411813 (N=12) | OLE: Cohort 1: JNJ-40411813 Followed by JNJ-40411813 (N=23) | OLE: Cohort 2: Placebo Followed by JNJ-40411813 (N=7) | OLE: Cohort 2: JNJ-40411813 Followed by JNJ-40411813 (N=31)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 5 | 0 | 1 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 4 | 0 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood Chloride Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 4 | 1 | 3 | 0 | 2
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 3 | 1 | 3 | 0 | 1 | 2 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04836559/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04836559/SAP_001.pdf